CLINICAL TRIAL: NCT01382771
Title: A Randomized, Double-Blind, Placebo Controlled Perspective Study of Intraarticular Lumbar Zygapophysial Joint Corticosteroid Injection(s) as a Treatment of Chronic Low Back Pain in a Selected Population
Brief Title: Intraarticular Lumbar Joint Corticosteroid Injection(s) as a Treatment of Chronic Low Back Pain in a Selected Population
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 319-2010
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Low Back Pain
Keywords: low back pain; zygapophysial joint pain; medial branch block; > 6 months duration; non-radicular
MeSH Terms: conditions — Low Back Pain | interventions — Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-articular corticosteroid injection (Active Comparator): Intra-articular corticosteroid injection in conjunction with confirmatory anesthetic medial branch blocks
  Interventions: Drug: Intra-articular corticosteroid injection
- Intra-articular saline injection (Placebo Comparator): Intra-articular saline injections with confirmatory anesthetic medial branch blocks
  Interventions: Drug: Intra-articular saline injection

INTERVENTIONS:
Drug: Intra-articular corticosteroid injection — Intra-articular injection of 0.5 cc triamcinolone acetonide (40 mg/cc) within each joint
  Arms: Intra-articular corticosteroid injection
Drug: Intra-articular saline injection — Intra-articular injection of 0.5 cc normal saline in each joint
  Arms: Intra-articular saline injection

SUMMARY:
Subjects (N=120) who have had non-radicular low back pain, believed by clinical assessment and imaging to be consistent with lumbar zygapophysial joint (Z-joint) generated pain, who have failed conservative therapy including physical therapy, have had an initial >80% pain relief on a diagnostic medial branch block, and are scheduled to undergo a routine second medial branch block for facet mediated pain will be randomized. Both groups will receive the standard of care, a medial branch block. The treatment group will also receive one set of intra-articular lumbar Z-joint corticosteroid injection and the placebo group will receive intra-articular normal saline.

DETAILED DESCRIPTION:
Subjects will have failed conservative treatment, including, but not limited to oral medications, physical therapy, chiropractic treatment, and/or alternative medicine. They will be evaluated by a spine specialist in the Spine Division of the Department of Orthopaedics and will be schedule for a medial branch block as standard of care. As part of usual and standard care, patients will undergo lumbar medial branch blocks for diagnosis of zygapophysial joint pain.

Patients who obtain ≥ to 80% relief of their index pain with a first set of lumbar medial branch blocks will be offered the opportunity for possible inclusion in the study if they are scheduled to receive a second medial branch block. The definition of a positive response to MBB's is an 80% reduction in pain (by change in NPR scores or estimated patient improvement) AND the restoration of the ability to perform at least one previously painful posture, movement, or activity without increase in pain, during the anesthetic phase of the blocks. If subjects are unable to render NPR scores or percentage estimate of improvement, then a 5 point global perception of effect tool will be used.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain episode greater than six months in duration
* NPR pain scale score three day average and present pain of at least four/ten at baseline (index pain)
* Previous medial branch block providing >80% pain relief for current painful episode
* Subject must be scheduled to undergo a second medial branch block for their back pain

Exclusion Criteria:

* Litigation
* Those seeking new or increased long-term remuneration
* Leg pain greater than back pain
* Radicular pain or evidence of neurological compromise in the lower limbs
* Those unable to read English and complete the assessment instruments
* Systemic inflammatory arthritis (e.g. rheumatoid, lupus)
* Addictive behavior, severe clinical depression or psychotic features. The subjects will be identified at the sole discretion of the PI who per the current standard of care will consent the potential subjects to the study
* Significant lower extremity pathology that affects gait
* Sustained cervical or thoracic pain that is present at a level >3/10 on NPR
* Possible pregnancy or other reason that precludes the use of fluoroscopy
* Significant scoliosis
* Radicular/neurological deficits or focal disc herniation and/or stenosis, with correlating radicular symptoms
* Contra-indication to corticosteroid, including known allergies or sensitivities
* History of prior epidural spinal injections relieving their current pain, or prior lumbar surgery.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating (NPR) or patient estimation of improvement, >80% pain reduction | Hourly for 6 hours post injections
  A positive response is defined as are ≥ 80% reduction in pain (by change in NPR scores or estimated patient improvement) AND the restoration of the ability to perform at least one previously painful posture, movement, or activity without increase in pain, during the anesthetic phase of the blocks.

SECONDARY OUTCOMES:
Numeric Pain Rating (NPR) Daily diary | reviewed at 6 weeks, 3 months, 6 months, 12 months follow-up
  The patient will be instructed to maintain a pain diary that records the degree and duration of any relief.
Oswestry Disability Index (ODI) | 6 weeks, 3 months, 6 months, 12 months
  Patient will complete ODI at the follow-up intervals.
Standard Form 36 (SF-36), General Health Survey | 6 weeks, 3 months, 6 months, 12 months
  Patient will complete the SF-36 at the follow-up intervals. The SF-36 is a self-administered, generic, general health survey consisting of 36 questions. The questions focus on the functional health and well being of the subject completing the form.
Daily Work History Log | reviewed at the 6 weeks, 3months, 6 months, 12 months follow-up
  Patient will keep a Work History Log during participation. The Log should indicate the daily work activities of the subject.
Daily Analgesic Use Log | reviewed at 6 weeks, 3 months, 6 months, 12 months
  Patient will keep a Daily Analgesic Use Log during participation.
Ancillary Treatment Log | reviewed at 6 weeks, 3 months, 6 months, 12 months follow-up
  Patient will keep an Ancillary Treatment Log during participation. This log will indicate any outside medical care, additional medial branch blocks or radiofrequency neurotomy treatments.

CONTACTS AND LOCATIONS:
Overall Officials: D. J. Kennedy, M.D., Principal Investigator — UF Department of Orthopaedics and Rehabilitation
Locations (1):
- UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States